CLINICAL TRIAL: NCT04663074
Title: Prospective Register of Anatomical / Geometric Data Obtained by Intravascular Ultrasound (IVUS) Examinatio´n of Bridging Stent Grafts in Complex Aortic Interventions
Brief Title: Intravascular Ultrasound (IVUS) in Complex Aortic Endovascular Interventions
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: 01_2020
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-05

CONDITIONS: Thoracic Aortic Aneurysm
Keywords: Intravascular ultrasound; bridging stentgraft; BEVAR; EVAR; IVUS
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IVUS Group: Patients treated by BEVAR/CHEVAR/FEVAR due to a thoracoabdominal aneurysm.
  Interventions: Diagnostic Test: IVUS control

INTERVENTIONS:
Diagnostic Test: IVUS control — Intravascular Control of the bridging stentgrafts during branched EVAR
  Other Names: Volcano Philips

SUMMARY:
The study aims to investigate the applicability of intravascular ultrasound (IVUS) in the endovascular therapy of juxta-, supra- and thoracoabdominal aortic aneurysms.

The focus of the study is on the intraoperative and postoperative evaluation of the geometric data of bridging stentgrafts in terms of patency, occurrence of stenosis and/or kinking.

DETAILED DESCRIPTION:
Intravascular ultrasound (IVUS) is an already validated diagnostic method increasingly use in endovascular interventions. In contrast to conventional digital subtraction angiography (DSA), the IVUS provides in vivo real-time vessel images. Furthermore, its accuracy has been examined in histological studies, which could report of a good correlation regarding the vessel diameters (Jin ZG et al. Int J Cardiovasc Imaging. 2017 Feb; 33 (2): 153-160.).

Stenosis and/or kinkings of stents or stentgrafts as well as their fully expansion and morphology can be assessed with the use of IVUS.

The IVUS has already been used successfully in the context of endovascular treatment of infrarenal aortic aneurysms (Endovascular Aortic Repair or EVAR). Here, the IVUS has proven to be a valuable diagnostic instrument to examine the anatomy of the inserted stent grafts intraoperatively and to detect any abnormalities. In addition, the use of IVUS led to a significant reduction in the use of iodine-containing contrast media and radiation exposure as part of these complex endovascular interventions (Pecoraro F et al. Ann Vasc Surg. 2019 Apr; 56: 209-215.).

In the endovascular therapy of thoracoabdominal as well as suprarenal and juxtarenal aortic aneurysms, stent grafts with recesses (windows - Fenestrated EVAR or FEVAR) or side arms (branches - Branched EVAR or BEVAR) for the renovisceral vessels (truncus coeliacus, superior mesenteric artery and renal arteries) are implanted. In exceptional cases, the renovisceral vessels are supplied with stent grafts that are implanted in parallel to the aortic stent grafts (Chimney-Technique). These branches or windows are then connected to the corresponding target vessels via a bridging stent graft. The patency and anatomy of the bridging stent grafts are usually checked intraoperatively by angiography. The dynamics of the contrast agent flow and the X-ray images of the framework of the stent graft help in assessing their patency as well as the absence of structural problems.

The Computed Tomographic Angiography (CTA) is considered the gold standard as diagnostic method to assess the patency and anatomy of the stentgrafts postoperatively. This diagnostic method bares with it the exposure to relevant radiation dose as well as to contrast media. However, CTA scans do not provide in vivo real-time vessel images.

Furthermore, in case of pathological findings a new intervention may be necessary. The IVUS technique overcomes these issues due to its low invasiveness and its possible use during the index procedure. This can lead to the immediate identification of eventual structural problems of the bridging stent grafts which can jeopardize their patency and to correct them already during the index procedure.

The use of the IVUS during FEVAR, BEVAR and CHEVAR has already been implemented in our clinical routine. At our knowledge, a prospective collection of anatomical-geometric data by IVUS in complex endovascular treatments of complex aortic aneurysm has not been yet reported.

The aim of the current study is the retrospective evaluation of the anatomical-geometric data already collected by IVUS as well as the prospective collection of new data regarding the patency and anatomy of bridging stent grafts.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Elective or emergency treatment of an aortic aneurysm with a branched or fenestrated stent graft or with the aid of parallel stent grafts´(chimney)
* Patient capable of giving informed consent

Exclusion Criteria:

* Patients who are already participating in another study
* child bearing or breast feeding females

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by BEVAR/CHEVAR/FEVAR due to a thoracoabdominal aneurysm,
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
bSG patency | 5 years
  Patency of the bridging stentgraft

SECONDARY OUTCOMES:
Geometrical changes | 5 years
  Geometrical changes of the bridging stentgrafts during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Oberhuber, Principal Investigator — University Hospital Muenster
Locations (6):
- Department of Vascular Surgery, Rigshopitalet, Copenhagen, Denmark
- Germany (2):
  - Klinik für Gefäßchirurgie, St. Franziskus-Hospital, Münster
  - Muenster University Hospital, Münster
- Italy (2):
  - Vascualar Surgery, Nocsae Nuovo Ospedale Civile di Baggiovara St. Agostiono Estense, Modena
  - Vascular and Endovascular Surgery Division, Padua University, Padua
- Division of Vascular Surgery, Uppsala University, Upplands Vasby, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jin ZG, Zhang ZQ, Jing LM, Wei YJ, Zhang J, Luo JP, Yang SL, Ma DX, Liu Y, Han W, Yang Y, Liu HL. Correlation between dual-axis rotational coronary angiography and intravascular ultrasound in a coronary lesion assessment. Int J Cardiovasc Imaging. 2017 Feb;33(2):153-160. doi: 10.1007/s10554-016-0999-5. Epub 2016 Oct 11. PMID 27730313
- [Background] Pecoraro F, Bracale UM, Farina A, Badalamenti G, Ferlito F, Lachat M, Dinoto E, Asti V, Bajardi G. Single-Center Experience and Preliminary Results of Intravascular Ultrasound in Endovascular Aneurysm Repair. Ann Vasc Surg. 2019 Apr;56:209-215. doi: 10.1016/j.avsg.2018.09.016. Epub 2018 Nov 27. PMID 30500656
- [Background] Georgiadis GS, van Herwaarden JA, Antoniou GA, Hazenberg CE, Giannoukas AD, Lazarides MK, Moll FL. Systematic Review of Off-the-Shelf or Physician-Modified Fenestrated and Branched Endografts. J Endovasc Ther. 2016 Feb;23(1):98-109. doi: 10.1177/1526602815611887. Epub 2015 Oct 23. PMID 26496957
- [Background] Mafeld S, Annamalai G, Lindsay TF, Zhong I, Tarulli E, Mironov O, Tan KT. Initial Experience With Viabahn VBX as the Bridging Stent Graft for Branched and Fenestrated Endovascular Aneurysm Repair. Vasc Endovascular Surg. 2019 Jul;53(5):395-400. doi: 10.1177/1538574419840880. Epub 2019 Apr 24. PMID 31018828
- [Background] Spear R, Sobocinski J, Hertault A, Delloye M, Azzauiu R, Fabre D, Haulon S. One Year Outcomes of 101 BeGraft Stent Grafts used as Bridging Stents in Fenestrated Endovascular Repairs. Eur J Vasc Endovasc Surg. 2018 Apr;55(4):504-510. doi: 10.1016/j.ejvs.2018.01.023. Epub 2018 Mar 1. PMID 29501401
- [Background] Donas KP, Lee JT, Lachat M, Torsello G, Veith FJ; PERICLES investigators. Collected world experience about the performance of the snorkel/chimney endovascular technique in the treatment of complex aortic pathologies: the PERICLES registry. Ann Surg. 2015 Sep;262(3):546-53; discussion 552-3. doi: 10.1097/SLA.0000000000001405. PMID 26258324
- [Background] Timaran DE, Knowles M, Soto-Gonzalez M, Modrall JG, Tsai S, Kirkwood M, Rectenwald J, Timaran CH. Gender and perioperative outcomes after fenestrated endovascular repair using custom-made and off-the-shelf devices. J Vasc Surg. 2016 Aug;64(2):267-272. doi: 10.1016/j.jvs.2016.02.062. Epub 2016 Jun 15. PMID 27316411
- [Background] Verhoeven EL, Katsargyris A, Oikonomou K, Kouvelos G, Renner H, Ritter W. Fenestrated Endovascular Aortic Aneurysm Repair as a First Line Treatment Option to Treat Short Necked, Juxtarenal, and Suprarenal Aneurysms. Eur J Vasc Endovasc Surg. 2016 Jun;51(6):775-81. doi: 10.1016/j.ejvs.2015.12.014. Epub 2016 Feb 6. PMID 26860255
- [Background] Mastracci TM, Carrell T, Constantinou J, Dias N, Martin-Gonzalez T, Katsargyris A, Modarai B, Resch T, Verhoeven EL, Burnell M, Haulon S. Editor's Choice - Effect of Branch Stent Choice on Branch-related Outcomes in Complex Aortic Repair. Eur J Vasc Endovasc Surg. 2016 Apr;51(4):536-42. doi: 10.1016/j.ejvs.2015.12.046. Epub 2016 Feb 23. PMID 26916389